CLINICAL TRIAL: NCT04982107
Title: Pupil Influence on the Quality of Vision in Implantable Collamer Lens (ICL)
Brief Title: Quality of Vision in Implantable Collamer Lens (ICL)
Status: Completed | Type: Observational
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ICL2020
Record Dates: First submitted 2021-01-26; First posted 2021-07-29 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-07

CONDITIONS: Pupil Diameter
Keywords: ICL; QoV; Visual acuity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to observe the influence of pupil size upon visual outcome in patients with Visian Implantable Collamer Lens(ICL) and toric-ICL implantation.

DETAILED DESCRIPTION:
The aim of this study is to observe the influence of pupil size upon the quality of vision outcome in patients with Visian Implantable Collamer Lens(ICL) and toric-ICL implantation. Pre-operation and 3-month post-operation pupil size, visual acuity, quality of vision will be evaluated in patient that had ICL surgery.

ELIGIBILITY:
Inclusion Criteria:

* Myopic eyes
* Preoperative corneal endothelial cell count ≥2200/mm2
* Preoperative central anterior chamber depth> 2.80mm
* Intraocular pressure within the normal range (10-21mmHg)

Exclusion Criteria:

* Severe dry eye
* Cataract and glaucoma
* Patients with uveitis
* Retinal detachment
* Patients with autoimmune diseases
* Patients with systemic diseases such as diabetes and hypertension
* Patients with mental or cognitive abnormalities

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Randomly choosen patients from the hospital records who had ICL surgery at He Eye Hospital, Shenyang, China during September 2019 to September 2020. They must have signed informed consent for their records to be used for education and research purposes before undergoing ICL surgery for myopic correction.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Subjective Quality of vision | Baseline (before surgery) and 3 month after surgery
  Change in QoV questionnaire score after ICL surgery at 3-month testing will be compare with baseline measurements
Pupil diameter pre-operation and post-operation | Baseline (before surgery) and 3 month after surgery
  Change in Pupil diameter after ICL surgery at 3-month testing will be compare with baseline measurements
Wave front aberrometry | baseline and 3 month after surgery
  Change in Wave front aberrometry after ICL surgery at 3-month testing will be compare with baseline measurements
Point Spread Function (PSF) | baseline and 3 month after surgery
  Change in Point Spread Function (PSF) after ICL surgery at 3-month testing will be compare with baseline measurements
Strehl ratio | Baseline and 3 month after surgery
  Change in Pupil diameter after ICL surgery at 3-month testing will be compare with baseline measurements
Modulation transfer function (MTF) | Baseline and 3 month after surgery
  Change in Modulation transfer function after ICL surgery at 3-month testing will be compare with baseline measurements

CONTACTS AND LOCATIONS:
Overall Officials: Wei He, Study Chair — He Eye Specialist Hospital, Shenyang.
Locations (1):
- He Eye Specialist Hospital, Shenyang., Shenyang, Liaoning, China